CLINICAL TRIAL: NCT01702025
Title: Rapid Acclimatization to Hypoxia at Altitude
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Defense Advanced Research Projects Agency (U.S. Federal Agency); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Christopher Bell, Associate Professor, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N66001-10-C-2134
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Physiological Function in Low Oxygen Environment
Keywords: Hypoxia; Altitude; Exercise
MeSH Terms: conditions — Hypoxia; Motor Activity | interventions — Aminophylline; Theophylline; Methazolamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Administer a single dose of placebo (yellow corn meal in a capsule, gelatin ) in Normoxic Conditions.
  Following a minimum of 7 days a single dose placebo will be administered (yellow corn meal in a gelatin capsule) in Hypoxic conditions.
  Interventions: Drug: Placebo
- Aminophylline (Active Comparator): Administer a single dose of 400 mg Aminophylline (4-100 mg tablets) in Normoxic Conditions.
  Following a minimum of 7 days administer a single dose of 400 mg Aminophylline (4-100 mg tablets) in Hypoxic conditions.
  Interventions: Drug: Aminophylline
- Methazolamide (Active Comparator): Administer a single dose of 250 mg Methazolamide (10-25 mg tablets) in Normoxic Conditions.
  Following a minimum of 7 days administer a single dose of 250 mg Methazolamide (10-25 mg tablets) in Hypoxic conditions.
  Interventions: Drug: Methazolamide
- Aminophylline+Methazolamide (Active Comparator): Administer a single dose of 400 mg Aminophylline (4-100 mg tablets) + 250 mg Methazolamide (10-25 mg tablets) in Normoxic Conditions.(Aminophylline+Methazolamide)
  Following a minimum of 7 days administer a single dose of 400 mg Aminophylline (4-100 mg tablets) + 250 mg Methazolamide (10-25 mg tablets) in Hypoxic conditions.
  Interventions: Drug: Aminophylline+Methazolamide

INTERVENTIONS:
Drug: Placebo — Yellow corn meal in gel capsules
  Other Names: Yellow corn meal
  Arms: Placebo
Drug: Aminophylline — National Drug Code (NDC) 0143-1020-01
  Other Names: Theophylline
  Arms: Aminophylline
Drug: Methazolamide — NDC 0781-1072-01
  Other Names: Neptazane
  Arms: Methazolamide
Drug: Aminophylline+Methazolamide — NDC 0143-1020-01 and NDC 0781-1072-01
  Other Names: Theophylline + Neptazane
  Arms: Aminophylline+Methazolamide

SUMMARY:
In low oxygen environments, such as altitude, some adults may become ill and suffer from acute mountain sickness. Further, all adults will find that exercising becomes much more difficult when compared with exercise at lower altitudes (e.g. sea-level). The purpose of this investigation is to study the effects of two drugs that may help people adjust to high-altitude quickly, prevent them from becoming ill and improve their exercise performance. The drugs are Methazolamide and Aminophylline.

ELIGIBILITY:
Inclusion Criteria:

* normotensive (i.e. <140/90 mmHg)

Exclusion Criteria:

* Pregnancy
* nursing mother
* current tobacco use or regular use within the previous two years
* use of prescription medication other than birth control
* asthma or any other type of lung/respiratory dysfunction
* resting oxygen saturation <95%
* unwillingness to abstain from exercise for 48 hours prior to laboratory testing
* use of anticoagulant therapy or have a known or suspected bleeding disorder
* identification of contraindication during screening (i.e. positive stress test)
* any history of mountain sickness (altitude sickness)
* any history of allergic reaction, hypersensitivity or idiosyncratic reaction to any of the products administered during the study, including allergy to any sulfa or sulfonamide derivatives
* history of clinically significant illness within 4 weeks prior to Day 1
* Subjects who have made any significant donation (including plasma) or have had a significant loss of blood within 30 days prior to visit 1
* receipt of a transfusion or any blood products within 30 days prior to visit 1.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bell, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Dept. of Health and Exercise Science, Fort Collins, Colorado, United States

REFERENCES:
- [Derived] Scalzo RL, Binns SE, Klochak AL, Giordano GR, Paris HL, Sevits KJ, Beals JW, Biela LM, Larson DG, Luckasen GJ, Irwin D, Schroeder T, Hamilton KL, Bell C. Methazolamide Plus Aminophylline Abrogates Hypoxia-Mediated Endurance Exercise Impairment. High Alt Med Biol. 2015 Dec;16(4):331-42. doi: 10.1089/ham.2015.0066. PMID 26680684
- See also: Department of Health and Exercise Science, Colorado State University — http://hes.chhs.colostate.edu/
- See also: Initial Safety Trial For Treatments Under Investigation In Current Study — http://clinicaltrials.gov/ct2/show/NCT01587027?term=THE+SAFETY+EVALUATION+OF+AMINOPHYLLINE+AND+METHAZOLAMIDE+WHEN+ADMINISTERED+ORALLY+ALONE+AND+IN+COMBINATION+TO+HEALTHY+VOLUNTEERS&rank=1

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 19 individual participants enrolled in the study. Participants were provided with the opportunity to re-enroll and enter additional arm(s).
Groups:
- Placebo: Single dose Placebo Normoxia Minimum 7 day washout Single dose placebo: Hypoxia
- Aminophylline: Single dose Aminophylline Normoxia Minimum 7 day washout Single dose Aminophylline Hypoxia
- Methazolamide: Single dose Methazolamide Normoxia Minimum 7 day washout Single dose Methazolamide: Hypoxia
- Aminophylline + Methazolamide: Single dose Aminophylline+Methazolamide Normoxia Minimum 7 day washout Single dose Aminophylline+Methazolamide: Hypoxia
Period: Overall Study
Arm/Group | Placebo | Aminophylline | Methazolamide | Aminophylline + Methazolamide
Started | 11 | 10 | 10 | 10
Completed | 9 | 9 | 9 | 10
Not Completed | 2 | 1 | 1 | 0
Not completed — Equipment failure | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects could choose to participate in multiple arms of the trial. Trial arms were separated by a 7 day wash out period following the hypoxia visit of the previous arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Aminophylline | Methazolamide | Aminophylline + Methazolamide | Total
Number analyzed (Participants) | 11 | 10 | 10 | 10 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 10 | 10 | 41
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (5) | 26 (7) | 27 (6) | 27 (5) | 27 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2 | 4
  Male | 10 | 9 | 10 | 8 | 37
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 10 | 10 | 41
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.8 (2) | 25.4 (2) | 25.1 (2) | 25.4 (2) | 25.2 (2)
Body Fat % [Mean (Standard Deviation); unit: Percentage of body fat] | 20.2 (3) | 21.4 (7) | 20.6 (2) | 22.4 (7) | 21.1 (5)
Fat Mass [Mean (Standard Deviation); unit: kilograms] | 15.4 (2) | 16.5 (5) | 16.0 (2) | 17.4 (5) | 16.3 (3)
Fat Free Mass [Mean (Standard Deviation); unit: kilograms] | 61.3 (7) | 60.8 (8) | 61.9 (7) | 60.9 (9) | 61.2 (7)
maximal oxygen uptake (VO2max) [Mean (Standard Deviation); unit: milliliter/kilogram/minute] | 48.7 (8) | 49.4 (10) | 49.8 (8) | 46.5 (8) | 48.6 (8)

OUTCOME MEASURES:

1. Primary Outcome: Magnitude of Decrement in Exercise Time Trial Performance in Hypoxia (Low Oxygen) Compared With Normoxia (Normal Oxygen).
Description: After exercising on a stationary cycle ergometer for 30 minutes at a resistance of 100 watts, research participants will complete an exercise time trial. The time taken to cycle a distance equivalent to 7.75 miles will be recorded. On a separate day the experiment will be repeated in hypoxia. It is expected that the time taken to cycle a distance equivalent to 7.75 miles will be longer in hypoxia compared to normoxia. One of the goals of this research is to determine if the hypoxia-mediated performance decrement can be decreased with one of our pharmacological interventions.
Time Frame: The exercise trial will begin within 5 hours of exposure to either normoxia or hypoxia
Measure: Mean (Standard Error); unit: minutes
Groups:
- Normoxia Placebo: Placebo: single dose Normoxia
- Hypoxia Placebo: Placebo: single dose hypoxia
- Normoxia Aminophylline: Aminophylline:single dose Normoxia
- Hypoxia Aminophylline: Aminophylline:single dose hypoxia
- Normoxia Methazolamide: Methazolamide single dose Normoxia
- Hypoxia Methazolamide: Methazolamide: single dose hypoxia
- Normoxia Methazolamide/Aminophylline: Methazolamide combined with Aminophylline: single dose normoxia
- Hypoxia Methazolamide/Aminophylline: Methazolamide combined with Aminophylline: single dose hypoxia
Arm/Group | Normoxia Placebo | Hypoxia Placebo | Normoxia Aminophylline | Hypoxia Aminophylline | Normoxia Methazolamide | Hypoxia Methazolamide | Normoxia Methazolamide/Aminophylline | Hypoxia Methazolamide/Aminophylline
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 10 | 10
minutes | 22.3 (0.7) | 25.2 (1.2) | 22.2 (0.5) | 24.0 (0.7) | 23.0 (0.5) | 24.6 (0.5) | 24.5 (0.9) | 25.9 (1.0)

ADVERSE EVENTS:
Groups:
- Placebo: Single dose Placebo Normoxia Minimum 7 day washout Single dose placebo Hypoxia
  .
- Methazolamide: Single dose Methazolamide Normoxia Minimum 7 day washout Single dose Methazolamide Hypoxia
Arm/Group | Placebo | Aminophylline | Methazolamide | Aminophylline + Methazolamide
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/11 | 1/10 | 2/10 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | Aminophylline (N=10) | Methazolamide (N=10) | Aminophylline + Methazolamide (N=10)
Face Tingling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) — Tingling sensation in the face
Double vision (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lightheadedness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasovagal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Vasovagal response following needle stick
Hypoglycemic event (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cardiac rhythm (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Changes in premature ventricular contraction 24 days post consumption of study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No